CLINICAL TRIAL: NCT03843398
Title: Survival Outcome After Minilaparotomy for the Treatment of Colorectal Cancer
Acronym: SoMiniCRC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, En-Da Yu, Director of Department of Colorectal Surgery and Vice Director of GI Endoscopy, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SINOCOLO2019C
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Minilaparotomy; Survival
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Laparotomy; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minilaparotomy Group (Experimental): Participants in this arm undergo colorectal cancer resection via minilaparotomy.
  Interventions: Procedure: Colorectal cancer resection via minilaparotomy
- Laparoscopy Group (Active Comparator): Participants in this arm undergo laparoscopic colorectal cancer resection.
  Interventions: Procedure: Laparoscopic colorectal cancer resection

INTERVENTIONS:
Procedure: Colorectal cancer resection via minilaparotomy — According to the cancer location, a 7 cm incision is made in specific area of the patient's abdomen. The whole procedure of operation will be finished within this incision. If the incision must be lengthen due to the surgical demand, the failure of the minilaparotomy is determined.
  Other Names: Minilaparotomy
  Arms: Minilaparotomy Group
Procedure: Laparoscopic colorectal cancer resection — This is one of the routine procedures used for colorectal cancer resection.
  Other Names: Laparoscopy
  Arms: Laparoscopy Group

SUMMARY:
The primary aim of this study is

- to determine the difference of survival outcome (3-year overall survival, 3y OS) between after minilaparotomy and after laparoscopy..

Other aims include to determine the data below when minilaparotomy and laparoscopy are compared with each other.

* 3-year disease free survival, 3y DFS
* 5-year overall survival, 5y OS
* 5-year disease free survival, 5y DFS
* Local recurrence rate, LRR
* Postoperative complications Incidence and mortality at 30 days

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer with pathological results.
* Colorectal cancer preliminary diagnosed during colonoscopy.
* No confirmed metastasis.
* No comorbidity of other malignancy.
* The primary tumor is less than 10 cm.
* No organ dysfunction.
* The patient and his families totally agree with the whole investigative procedure, and sign the written informed consent form.

Exclusion Criteria:

* Diagnosed with any other malignancy within 5 years.
* Comorbidity of emergent conditions like perforation.
* Former colorectal surgery history which may affects digestive tract reconstruction.
* Need combined organ resection.
* ASA grade IV or V.
* Pregnant or lactating Women.
* Severe mental diseases.
* Severe cardiopulmonary diseases which reduce operation tolerance.
* Systematic steroid therapy lasting for more than 1 month.
* Intolerant of laparoscopy.
* No written informed consent form signed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival, 3y OS | 3 years after the follow up of the last patient enrolled.
  3y OS

SECONDARY OUTCOMES:
5-year overall survival, 5y OS | 5 years after the follow up of the last patient enrolled.
  5y OS
3-year disease free survival, 3y DFS | 3 years after the follow up of the last patient enrolled.
  3y DFS
5-year disease free survival, 3y DFS | 5 years after the follow up of the last patient enrolled.
  5y DFS
Local recurrence rate, LRR | 3 years after the follow up of the last patient enrolled.
  LRR
Postoperative complications Incidence at 30 days | 30 days after the operation of the last patient enrolled.
  PCI30
Postoperative mortality at 30 days | 30 days after the operation of the last patient enrolled.
  PM30

CONTACTS AND LOCATIONS:
Overall Officials: En-Da YU, MBBS, Principal Investigator — Changhai Hospital

REFERENCES:
- [Background] Wang XD, Huang MJ, Yang CH, Li K, Li L. Minilaparotomy to rectal cancer has higher overall survival rate and earlier short-term recovery. World J Gastroenterol. 2012 Oct 7;18(37):5289-94. doi: 10.3748/wjg.v18.i37.5289. PMID 23066325
- [Background] Ishida H, Ishiguro T, Ohsawa T, Okada N, Kumamoto K, Ishibashi K, Haga N, Yokoyama M, Nakada H, Gonda T. Oncologic outcome of stages II/III colon cancer treated via minilaparotomy. Int Surg. 2011 Apr-Jun;96(2):127-34. doi: 10.9738/1384.1. PMID 22026303
- See also: PubMed link — http://www.ncbi.nlm.nih.gov/pubmed/23066325
- See also: PubMed link — http://www.ncbi.nlm.nih.gov/pubmed/22026303